CLINICAL TRIAL: NCT03356483
Title: Psilocybin Treatment in Obsessive-Compulsive Disorder: a Preliminary Efficacy Study and Exploratory Investigation of Neural Correlates.
Brief Title: Efficacy of Psilocybin in OCD: a Double-Blind, Placebo-Controlled Study.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Heffter Research Institute (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Benjamin Kelmendi, MD, Associate Research Scientist, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000020355; 1K23MH122777-01A1 (NIH)
Record Dates: First submitted 2017-11-06; First posted 2017-11-29 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Psilocybin
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Psilocybin; Niacin

STUDY DESIGN:
Intervention Model Description: In the study, half of the participants will be randomized to receive psilocybin (n=15) or the active-placebo-control, niacin (n=15). Following the first treatment session of either the active agent or active-placebo-control, participants who were randomized to receive active-placebo-control will be offered the option to receive open-label psilocybin. The blind will be broken at 48-hours to make this determination.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psilocybin (Experimental): Psilocybin (0.25mg/kg)
  Interventions: Drug: Psilocybin (0.25mg/kg)
- Niacin (Placebo Comparator): Niacin (250mg)
  Interventions: Drug: Niacin (250mg)

INTERVENTIONS:
Drug: Psilocybin (0.25mg/kg) — Psilocybin is a naturally occurring hallucinogenic ingredient found in some varieties of mushrooms that can be produced synthetically. It is considered to be a serotonergic psychedelic.
  Other Names: "Magic Mushrooms"
  Arms: Psilocybin
Drug: Niacin (250mg) — A medication used to treat high cholesterol, triglyceride levels, and niacin deficiency.
  Other Names: Nicotinic acid
  Arms: Niacin

SUMMARY:
This study aims to investigate the effects of oral psilocybin on OCD symptomatology and provide the first evidence of the neural mechanism that may mediate psilocybin's purported therapeutic effects on OCD.

DETAILED DESCRIPTION:
Aim 1: To investigate the effects of psilocybin on OCD symptomatology. OCD symptom severity will be assessed before treatment and 24 and 48 hours after treatment, one week after treatment, two weeks, one month, and three months after treatment. Hypothesis: We hypothesize that 0.25mg/kg of psilocybin will lead to greater symptom improvement than niacin (as the active-placebo-control agent) at the primary endpoint of 48 hours post-dosing and at all other assessment points.

Aim 2: To explore the relationship between the psilocybin-induced brain connectivity changes and symptom change in OCD. Resting-state brain connectivity will be assessed before and 48 hours after treatment. Hypothesis: We hypothesize that (i) psilocybin will normalize abnormal fronto-striatal functional connectivity in patients with OCD; and (ii) normalization of these abnormalities will correlate with improvement in symptomatology after psilocybin treatment.

This study will pilot a single-center, randomized, active-placebo-controlled, double-blind design to examine the clinical and neural effects on OCD, of either 0.25mg/kg of psilocybin or active placebo-control agent (niacin 250mg), given along with non-drug preparatory and follow-up support appointments to 30 study participants. The duration of the randomized study phase is from consent until two weeks after drug administration. Participants will be followed for 12 weeks (3 months) post-study drug administration.

Eligible participants will be admitted as an inpatient for at least 3 nights / 4 days surrounding the initial drug administration (or more, at the option of the subject and the investigator). Participants will be randomized into active medication and active-placebo-control groups, and will be blinded as to their study condition. This admission 2 nights prior to the drug administration will allow the participant to adjust to sleeping on the unit and allow them to settle in to the research unit routine. A return for an fMRI scan (48 hours after the administration session) will be scheduled. The participants who received active-placebo-control will be offered the option to receive open-label psilocybin.

ELIGIBILITY:
Inclusion Criteria:

1. Primary DSM-5 diagnosis of OCD
2. Y-BOCS score of 19 or greater
3. Failure of at least one trial of standard care treatment (medication and/or psychotherapy [CBT/ERP]) for OCD
4. English proficiency and fluency, and ability to understand the consent process and provide written informed consent
5. Willingness to sign a medical release for direct communication between research staff and external provider(s) about the participant's treatment and medical histories
6. Non-consumption of SSRIs for at least 8 weeks at the time of randomization
7. Willingness to refrain from psychiatric medications (e.g., antidepressants, first- and second-generation antipsychotics, mood stabilizers) during the study period, as well as certain other medications (e.g., anti-seizure medications, cardiovascular medications, and aldomet specifically) during the day of dosing
8. Willingness to abstain from THC-containing products for study duration. A negative urinary drug screen is also required at baseline and the day of dosing.
9. A negative urinary pregnancy screen at study entry and day of dosing if of childbearing potential, and willingness to use adequate birth control for study duration
10. Having a contact person who is willing and able to be reached by the study team in the event of an emergency/crisis, and who is able to transport the participant home at the end of the inpatient stay/dosing week
11. Willingness to commit to all study procedures and visits, including inpatient stay, assessments and self-reports, neuroimaging, and being medically cleared to be discharged and transported home at the end of the dosing week

Exclusion Criteria:

1. Personal or immediate family history of schizophrenia spectrum and other psychotic disorders, bipolar I or II disorder, or major depressive disorder with psychotic features
2. Active suicidal intent
3. Unremitted Tourette syndrome
4. Autism spectrum disorder
5. OCPD or BPD
6. Current substance use disorder (except mild alcohol use disorder)
7. Unstable neurological or medical condition(s) that may render study procedures unsafe, including poorly managed diabetes, hypertension, or cardiovascular conditions, or history of seizure(s) or chronic/severe headaches
8. Any history of head injury with loss of consciousness for more than 30 minutes
9. Any contraindications to undergoing an MRI scan, including having metal implants or metal fragments in the body
10. Any use of psychedelic substances within the prior 12 months

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Changes in severity of OCD symptoms, which will be measured by The Yale-Brown Obsessive-Compulsive Scale (Y-BOCS). The Primary Outcome Measure will be collected at baseline and 48 hours, assessing change from baseline at 48 hours. | Baseline, 48 hours post-drug, weeks: 1, 2, 4, 12 post-drug
  Assesses severity and types of OCD symptoms over the past seven days. Consists of two parts: 1- symptom checklist, 2- symptom severity scale. The most prominent obsessions and compulsions are identified by the checklist and then rated by the symptom severity scale. The symptom severity scale consists of 11 items (3 items are not included in the total score) and uses a 0 to 4 severity scale. Total Y-BOCS scores range from 0 to 40, with higher scores indicating greater severity of OCD symptoms.
Changes in severity of OCD symptoms, measured by Acute Yale-Brown Obsessive-Compulsive Scale (A-YBOCS) | Baseline, 24 hours post-drug, 48 hours post-drug
  A clinician-administered measure of specific participant OCD symptoms over prior 24 hours. The most prominent obsessions and compulsions that were previously identified by the checklist are rated by the symptom severity scale. The symptom severity scale consists of 11 items (3 items are not included in the total score) and uses a 0 to 4 severity scale. Total A-YBOCS scores range from 0 to 40, with higher scores indicating greater severity of OCD symptoms.
Changes in severity of OCD symptoms, measured by Visual Analog Scale (VAS) for OCD symptoms | Baseline, 24 hours post-drug, 48 hours post-drug
  A self-report measure of severity of and distress related to OCD symptoms over the past 24 hours. Consists of 5 items assessing compulsive urges, obsessions, anxiety, mood, and discomfort, each on a 0-100 VAS, with higher scores on each item indicating greater severity.
Changes in suicidality, measured by the Columbia-Suicide Severity Rating Scale (C-SSRS) Since Last Visit version | Up to 12 weeks post-drug
  A clinician-administered measure of suicidality since the last visit. Consists of 5 items assessing suicidal ideation and 6 items assessing suicidal and non-suicidal self-injurious behaviors. Higher scores on either scale indicate more severe suicidal ideation and suicidal or non-suicidal behaviors since the last study visit.

SECONDARY OUTCOMES:
Changes in brain connectivity, which will be measured with functional Magnetic Imaging Resonance (fMRI). | Baseline & 48 hours post-drug
  Resting-state brain connectivity will be assessed before and 48 hours after treatment. Neuronal activation induced by OCD-relevant provocative stimuli will be assessed 48 hours after the treatment.
Changes in depression symptoms, which will be measured by The Montgomery-Asberg Depression Scale (MADRS). | Baseline, 2 days post-drug, weeks: 1, 2, 4, 12, post-drug
  Assesses depression symptoms. Consists of 10 items and uses a 0 to 6 severity scale. Total scores range from 0 to 60, with higher scores indicating more severe depression.
Changes in depression symptoms, which will be measured by the Beck Depression Inventory (BDI). | Baseline, 1 day post-drug, weeks: 2 & 12 post-drug
  Assesses depression symptoms. Consists of 21 items and uses a 0 to 3 severity scale. Total scores range from 0 to 63, with higher scores indicating more severe depression.
Changes in dysfunctional beliefs, which will be measured by The Obsessive Beliefs Questionnaire (OBQ-44). | Baseline & 2 weeks post-drug
  Measures dysfunctional beliefs in obsessive-compulsive disorder. Consists of 44 items that are rated on a seven-point Likert scale, ranging from 1 (disagree very much) to 7 (agree very much). It contains three subscales: overestimations of threat and responsibility for harm (RT subscale), importance and control of intrusive thoughts (ICT subscale), and perfectionism and the need for certainty (PC subscale), with higher scores indicating higher levels of each sub-scale.
Changes in OCD symptoms, which will be measured by The Obsessive-Compulsive Inventory - Revised (OCI-R). | Baseline & 2 weeks post-drug
  An inventory of OCD symptoms. Consist of 18 items that are rated on a 5-point Likert scale. Total scores range from 0 to 72, with higher scores indicating more severe OCD symptoms.
Changes in OCD dimensions, which will be measured by The Obsessive-Compulsive Trait Core Dimensions Questionnaire (OC-TCDQ). | Baseline & 2 weeks post-drug
  Measures different OCD dimensions. Consists of 20 items assessing two core dimensions of OCD: harm avoidance (10 items) and incompleteness (10 items). Each item is rated from 0: never applies to me to 4: always applies to me. Higher scores on questions assessing harm avoidance indicates greater levels of harm avoidance. Higher scores on questions assessing incompleteness indicates higher levels of incompleteness.
Changes in anxiety, which will be measured by State-Trait Anxiety Inventory (STAI). | Baseline, 2 days post-drug, weeks: 1, 2, 4, 12 post-drug
  Measures state and trait anxiety. Consist of 40 items: 20 items measuring S-Anxiey and 20 items measuring T-Anxiety. State Anxiety Scale (S-Anxiety) evaluates the current state of anxiety. The Trait Anxiety Scale (T-Anxiety) evaluates relatively stable aspects of anxiety. The S-Anxiety scale assesses the intensity of current feelings "at this moment" from 1(not at all) to 4 (very much so). The T-Anxiety scale assesses the frequency of feelings "in general" from 1 (almost never) to 4 (almost always). The range of scores for each subtest is 20-80, with higher scores indicating greater anxiety.
Changes in quality of life, which will be measured by The Quality of Life Enjoyment & Satisfaction Questionnaire (Q-LESQ-SF). | Baseline, weeks: 2 & 12 post-drug
  Assesses quality of life and functionality. Consists of 16 items which are rated from 1 (very poor) to 5 (very good). Total score involves summing only the first 14 items to yield a raw total score. The raw total score ranges from 14 to 70. The raw total score is transformed into a percentage, with higher percentages indicating greater quality of life.
Changes in experiential aspects of psilocybin, which will be measured by The Mystical Experience Questionnaire (MEQ). | Day of drug administration, weeks: 2 & 12 post-drug
  Assesses different experiential aspects of psilocybin. Consists of 44 items which provides scale scores for each of seven domains of mystical experiences: Internal Unity (6 items); External Unity (6 items); Transcendence of Time and Space (8 items); Ineffability and Paradoxicality (5 items); Sense of Sacredness (7 items); Noetic Quality (4 items). Participants are asked to look back on the extended session that they have just experienced and to rate the degree of their experience of the following phenomena. Each item is rated from 0 (none; not at all) to 5 (extreme; more than ever before in my life and stronger than 4). Total scores are expressed as a proportion of the maximum possible score.
Changes in meaning of life, which will be measured by The Schedule for Meaning in Life Evaluation (SMiLE). | Baseline, weeks: 1 & 12 post-drug
  Assesses individual meaning in life. Participants are asked to name up to seven domains that they judge to be important to their individual meaning in life.Then they will rate their current level of satisfaction in each of these domains using a seven-point Likert scale (range, -3 to +3) and rate the importance of each of their chosen areas using a eight-point adjectival scale (range, 0 to 7). Higher total score indicate a greater meaning in life.
Challenging Experience Questionnaire (CEQ) | Day of drug administration
  Assesses difficult experiences induced by the interventions. Consists of 26 items that are rated from 0 (none; not at all) to 5 (extreme; more than ever before in my life). Participants are asked to rate the degree to which at any time during the previous session they experienced the following phenomena. Items are grouped into the following subscales: fear, grief, physical distress, insanity, isolation, death, and paranoia. Scores of each item are transformed into a percentage of the highest possible score. Subscale scores are calculated by averaging the transformed scores of the items in each subscale. The total score is the average of all the transformed item scores, with higher scores indicating more challenging experiences.
5-Dimension - Altered States of Consciousness (5D-ASC) | Day of drug administration
  Assesses different mental states induced by the interventions. Consists of 94 items which are rated by placing marks on a horizontal visual analogue scale (100 millimeters in length). The scale ranges from no, not more than usual (on the left) to yes, very much more than usual (on the right). The items are scored by measuring the millimeters from the low end of the scale to the participant's mark (from 0 to 100).
Changes in different dimensions of emotional experience, which will be measured by The Positive and Negative Affect Schedule Expanded Form (PANAS-X). | Baseline, 2 days post-drug, weeks: 1, 2, 4, 12 post-drug
  Assesses different dimensions of the emotional experience. This scale consists of 60 words and phrases that describe different feelings and emotions. For each item participants rate to what extent they have felt this way during the past few weeks from 1 (very slightly or not at all) to 5 (extremely). The items are grouped into the following 4 subgroups and subscales; general dimension scales (negative affect, positive affect), basic negative emotion scales (fear, hostility, guilt, sadness), basic positive emotion scales (joviality, self-assurance, attentiveness), other affective states (shyness, fatigue, serenity, surprise). The items pertaining to each subscale are summed with higher scores indicating higher levels of each subscale.
Changes of the effects of Psilocybin, which will be measured by The Persisting Effects Questionnaire (PEQ). | 2 days post-drug, weeks: 4 & 12 post-drug
  Assesses effects of Psilocybin. Consists of 86 items that assess eight categories of possible change in attitudes, mood, social effects, and behavior: 1. positive attitudes about life and/or self (17 items); 2. negative attitudes about life and/or self (17 items); 3. positive mood changes (4 items); 4. negative mood changes (4 items); 5. altruistic/positive social effects (8 items); 6. antisocial/negative social effects (8 items); 7. positive behavior changes (1 item); and 8. negative behavior changes (1item). Each item is rated using a 6-point rating scale from 0 (none, not at all) to 5 (extreme). Higher scores of each subscale indicate greater changes in that category.
Changes in connection to nature, which will be measured by The Nature Relatedness Scale (NRS). | Baseline & 2 weeks post-drug
  Assesses the affective, cognitive, and experiential aspects of individuals' connection to nature. Consists of 21 items which are rated on a 7-point Likert scale. The total score is calculated by averaging all 21 items after the appropriate items are reversed scored. Higher score indicate a greater connection with nature.
Changes in opinion towards pro-environmental behavior, which will be measured by The Pro-Environmental Behavior Scale (PEBS). | Baseline & 2 weeks post-drug
  Assesses opinions towards the importance of pro-environmental behaviors. Consists of 17 items that are rated from 1(not at all important) to 7 (extremely important). Higher total scores indicate a greater level of importance of pro-environmental behaviors.
Changes in anthropomorphism, which will be measured by The Individual Differences in Anthropomorphism Questionnaire (IDAQ). | Baseline & 2 weeks post-drug
  Assesses individual differences in anthropomorphism. Consists of 15 items which are rated by a 10-point Likert scale. Higher total scores indicate a higher level of anthropomorphism.
Changes in beliefs of mind-body dualism, which will be measured by The Mind-Body Dualism Scale (MBDS). | Baseline & 2 weeks post-drug
  Assesses beliefs of mind-body dualism. Consists of 11 items that are rated on a 7-point Likert scale. The total score is calculated after the appropriate items are reversed scored. Higher scores indicate a greater belief in mind-body dualism.
Change in interpersonal connectedness, which will be measured by The Inclusion of Others in Self Scale (IOS). | Baseline & 2 weeks post-drug
  Measures perceived interpersonal connectedness. A single-item, pictorial measure of closeness. Images range from the self and other as completely separate to the self and other almost completely overlapping.
Change in moral relativism and idealism, which will be measured by The Ethical Positions Questionnaire (EPQ). | Baseline & 2 weeks post-drug
  Assesses moral relativism and idealism. Consists of 20 items that are rated using a 9-point Likert scale (completely disagree to completely agree). Idealism scores are calculated by summing responses from items 1 to 10. Relativism scores are calculated by summing responses from items 11 to 20. Higher scores on items 1 to 10 indicate higher relativism and higher scores on items 11 to 20 higher idealism.
Changes in alcohol consumption, which will be measured by The Alcohol Use Disorders Identification Test (AUDIT). | Baseline & 12 weeks post-drug
  Assesses alcohol consumption, drinking behaviors, and alcohol-related problems. Consists of 10 items. The total score is calculated by summing all items. Higher scores indicate higher alcohol consumption. A score of 8 or more is considered to indicate hazardous or harmful alcohol use.
Changes in urgent care and emergency room use, which will be measured by The Utilization of Facility and Emergent Care (UFEC). | Baseline & 12 weeks post-drug
  Assesses frequency of urgent care and emergency room use. Consists of 26 items and 7 scales which include: Hypertension, High Cholesterol, Diabetes, Autoimmune, Musculoskeletal, Emergency Room Utilization, Urgent Care Utilization, Hospital Utilization, Facility Based Mental Health Care Utilization, Non-facility Based Mental Health Care Utilization. Items in each scale are scored by comparing follow-up scores to baseline scores. Positive difference indicates improved condition severity (Hypertension, High Cholesterol, Diabetes, Autoimmune, Musculoskeletal). Positive difference indicates reduced Emergency Room Utilization, Urgent Care Utilization, Hospital Utilization, Facility Based Mental Health Care Utilization, Non-facility Based Mental Health Care Utilization.
Changes in drug-related problems, which will be measured by The Drug Use Disorders Identification Test (DUDIT). | Baseline & 12 weeks post-drug
  Assesses drug-related problems. Consists of 11 items. The total score is calculated by summing all items. Drug related problems are indicated with a score of 6 or more for men and a score of 2 or more for women.
Changes in tobacco use, motivation to quit, and dependence, which will be measured by The Self-reported Nicotine Use (SRNU). | Baseline & 12 weeks post-drug
  Assesses tobacco use, motivation to quit, and dependence. Consists of 13 items. The baseline score of each item is compared to the follow-up score to assess changes. Higher scores indicate greater nicotine use.
Changes in sleep quality, which will be measured by The Pittsburgh Sleep Quality Index (PSQI). | Baseline, 48 hours post-drug, weeks: 4 & 12 post-drug
  Assesses sleep quality. Consists of 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available). Only self-rated questions are included in the scoring. The 19 self-rated items are combined to form seven "component" scores, each of which has a range of 0-3 points. In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The seven component scores are then added to yield one "global" score, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties in all areas.
Changes in readiness to change, which will be measured by The University of Rhode Island Change Assessment (URICA). | Baseline, 48 hours post-drug, weeks: 4, 8, 12 post-drug
  Assesses readiness to change. Consists of 30 items rated from 1(strongly disagree ) to 5 (strongly agree). Subscales include: Precontemplation, Contemplation, Action, and Maintenance. Subscale scores are calculated by averaging the items in each subscale. The total score is calculated by summing the subscales Contemplation, Action, Maintenance and subtracting Precontemplation. Higher score indicate greater readiness to change.
Changes in symptom severity and treatment response, which will be measured by The Clinical Global Impressions (CGI). | Baseline & 12 weeks post-drug
  Assesses symptom severity and treatment response. Consists of 4 items that are rated on a 7-point Likert scale. Symptom severity scores range from 1 (normal) through to 7 (amongst the most severely ill patients). Treatment response scores range from 1 (very much improved) through to 7 (very much worse). Each component is rated separately; this measure does not yield a global score. Higher scores indicate greater symptom severity and lower treatment response.
Changes in functional impairment, which will be measured by The Sheehan Disability Scale (SDS). | Baseline & 12 weeks post-drug
  Assesses functional impairment in three inter-related domains; work/school, social and family life. Impairment of each domain is rated from 0 (not at all) to 10 (extremely). The 3 items are summed into a single dimensional measure of global functional impairment that rages from 0 (unimpaired) to 30 (highly impaired).
Changes in optimism and pessimism, which will be measured by The Life Orientation Test Revised (LOT-R). | Baseline & 12 weeks post-drug
  Assesses individual differences in generalized optimism versus pessimism. Consists of 10 items that are rated from 0 (I agree a lot) to 4 (I disagree a lot). Of the 10 items, 3 items measure optimism, 3 items measure pessimism, and 4 items serve as fillers. Total scores are calculated by summing all items for a total ranging from 0 to 24.There are no "cut-offs" for optimism or pessimism; this measure is used as a continuous dimension of variability.
Changes in OCD symptoms, which will be measured by The Padua Inventory of OCD symptoms. | Baseline & 12 weeks post-drug
  Assesses OCD symptoms across five dimensions: (1) obsessional thoughts about harm to oneself or others; (2) obsessional impulses to harm oneself or others; (3) contamination obsessions and washing compulsions; (4) checking compulsions; and (5) dressing/grooming compulsions. Consists of 39 items that are rated from 0 (not at all) to 4 (very much). Items within each domain are summed for subscale scores. All items are summed for a total score with higher scores indicating greater symptom severity.
Changes in action identification, measured by the Behavior Identification Form (BIF) | Baseline & 1 week post-drug
  Assesses individual variation in identification of several motor actions and activities. Comprises 25 items of various motor actions or activities, of which each can be endorsed and interpreted on a binary response scale as either a literal motor action or a meaningful outcome-oriented behavior. Greater number of items responded literally or meaningfully indicate more literal or meaningful, outcome-oriented behaviors, respectively.
Changes in reactions to research participation, measured by the Reactions to Research Participation Questionnaire (RRPQ) | 48 hours post-drug and 12 weeks post-drug
  Assesses reactions to research participation. Consists of 26 items (each rated from 1-5) assessing various aspects of participation-related reactions, which can be parsed into 5 subscales: perceptions of participation, personal benefits, emotional reactions, perceived drawbacks, and global evaluation. Higher subscale scores indicate greater extent of respective reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Kelmendi, MD, Principal Investigator — Yale University; Christopher Pittenger, MD, PhD, Study Director — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moreno FA, Wiegand CB, Taitano EK, Delgado PL. Safety, tolerability, and efficacy of psilocybin in 9 patients with obsessive-compulsive disorder. J Clin Psychiatry. 2006 Nov;67(11):1735-40. doi: 10.4088/jcp.v67n1110. PMID 17196053
- [Background] Ross S, Bossis A, Guss J, Agin-Liebes G, Malone T, Cohen B, Mennenga SE, Belser A, Kalliontzi K, Babb J, Su Z, Corby P, Schmidt BL. Rapid and sustained symptom reduction following psilocybin treatment for anxiety and depression in patients with life-threatening cancer: a randomized controlled trial. J Psychopharmacol. 2016 Dec;30(12):1165-1180. doi: 10.1177/0269881116675512. PMID 27909164
- [Background] Griffiths RR, Johnson MW, Carducci MA, Umbricht A, Richards WA, Richards BD, Cosimano MP, Klinedinst MA. Psilocybin produces substantial and sustained decreases in depression and anxiety in patients with life-threatening cancer: A randomized double-blind trial. J Psychopharmacol. 2016 Dec;30(12):1181-1197. doi: 10.1177/0269881116675513. PMID 27909165
- [Background] Carhart-Harris RL, Erritzoe D, Williams T, Stone JM, Reed LJ, Colasanti A, Tyacke RJ, Leech R, Malizia AL, Murphy K, Hobden P, Evans J, Feilding A, Wise RG, Nutt DJ. Neural correlates of the psychedelic state as determined by fMRI studies with psilocybin. Proc Natl Acad Sci U S A. 2012 Feb 7;109(6):2138-43. doi: 10.1073/pnas.1119598109. Epub 2012 Jan 23. PMID 22308440
- [Derived] Ching THW, Grazioplene R, Bohner C, Kichuk SA, DePalmer G, D'Amico E, Eilbott J, Jankovsky A, Burke M, Hokanson J, Martins B, Witherow C, Patel P, Amoroso L, Schaer H, Pittenger C, Kelmendi B. Safety, tolerability, and clinical and neural effects of single-dose psilocybin in obsessive-compulsive disorder: protocol for a randomized, double-blind, placebo-controlled, non-crossover trial. Front Psychiatry. 2023 Apr 25;14:1178529. doi: 10.3389/fpsyt.2023.1178529. eCollection 2023. PMID 37181888